CLINICAL TRIAL: NCT02173275
Title: Computed TomogRaphic Evaluation of Atherosclerotic DEtermiNants of Myocardial IsChEmia (The CREDENCE Trial)
Brief Title: Computed TomogRaphic Evaluation of Atherosclerotic DEtermiNants of Myocardial IsChEmia
Acronym: CREDENCE
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1309014313; R01HL118019 (NIH)
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- derivation cohort: n = 309
- validation cohort: n = 309

SUMMARY:
The study seeks to determine the accuracy of using anatomic and physiologic information measurable by computed tomography features of stenosis, plaque, fractional flow reserve-CT and to compare this measure to stress testing for the detection of myocardial ischemia against the gold standard of cardiac catheterization with fractional flow reserve. The hypothesis of this proposal is that integrating anatomic plaque features with physiologic fractional flow reserve-CT will optimize identification of coronary lesions that are ischemia-causing by computed tomography .

DETAILED DESCRIPTION:
The CREDENCE trial will be a prospective multicenter cross-sectional study of 618 individuals (n=309 [derivation cohort]; n=309 [validation cohort]) who will undergo stress test, computed tomography, cardiac catheterization and fractional flow reserve. For the purposes of the study, either stress test or computed tomography will have been performed for clinical purposes, with the other test being performed as part of trial procedure. Study analyses will focus on the diagnostic performance of the information derived by stress test versus computed tomography against an invasive gold standard of cardiac catheterization and fractional flow reserve for an endpoint of vessel territory-specific ischemia. In keeping with prior studies, vessel territories will be comprised of the left anterior descending artery (and diagonal branches), the left circumflex artery (and obtuse marginal branches) and the right coronary artery (and posterolateral branch and posterior descending artery).

To date, the relative performance of traditional stress imaging testing compared to the entirety of information proffered by CT has not been assessed compared to an unbiased gold standard. The study proposed herein will directly address this unmet need.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Scheduled to undergo clinically-indicated non-emergent invasive coronary angiography

Exclusion Criteria:

1. Known CAD (myocardial infarction [MI], percutaneous coronary interventions [PCIs], coronary artery bypass graft [CABG],)
2. Hemodynamic instability
3. Inability to provide written informed consent
4. Concomitant participation in another clinical trial in which subject is subject to investigational drug or device
5. Pregnant state
6. Absolute contraindication to iodinated contrast due to prior near-fatal anaphylactoid reaction (laryngospasm, bronchospasm, cardiorespiratory collapse, or equivalent)
7. Serum creatinine ≥1.7 mg/dl or Glomerular Filtration Rate <30 ml/min
8. Baseline irregular heart rhythm (e.g., atrial fibrillation, etc.)
9. Heart rate ≥100 beats per minute
10. Systolic blood pressure ≤90 mm Hg
11. Contraindications to β blockers or nitroglycerin or adenosine
12. BMI >40 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive consenting adult patients who meet all of the inclusion criteria and none of the exclusion criteria will be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 618 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of vessel territory-specific ischemia of an integrated stenosis-APC-FFRCT measure by CT | 48-60 months
  The primary endpoint is the diagnostic accuracy of an integrated stenosis-APC-FFRCT metric by CT, as compared to perfusion or perfusion-MBF stress imaging testing for vessel territory-specific ischemia as determined by FFR (gold standard).

SECONDARY OUTCOMES:
Individual comparisons of APCs or FFRCT to MPI vessel-specific perfusion deficits or reduced MBF. | 48-60 months
  To compare the accuracy of the individual components of APCs or FFRCT to MPI vessel-specific perfusion deficits or reduced MBF against ischemia by FFR.
Post-PCI FFR prediction by FFRCT "virtual stenting" | 48-60 months
  To determine the accuracy of FFRCT "virtual stenting" to post-PCI FFR value of >0.80 and determine the correlation between the FFRCT "virtual stenting" to post-PCI FFR.

CONTACTS AND LOCATIONS:
Overall Officials: Leslee J Shaw, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (18):
- United States (10):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Mobile Cardiology Associates, Mobile, Alabama
  - Kaiser Permanente Hospital, San Jose, California
  - Oconee Heart and Vascular Center at St Mary's Hospital, Athens, Georgia
  - St. Luke's Lipid and Diabetes Research Center, Kansas City, Missouri
  - Renown Heart and Vascular, Reno, Nevada
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Hospital, Houston, Texas
  - Cardiac Center of Texas, McKinney, Texas
  - Multicare HS Institute for Research & Innovation, Tacoma, Washington
- Providence Health Care- St. Paul's Hospital; University of British Columbia, Vancouver, British Columbia, Canada
- State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China
- Italy (2):
  - Centro Cardiologico Monzino, IRCCS and University of Milan, Milan
  - Fondazione Toscana Gabriele Monasterio, Pisa
- St. Luke's Hospital, Tokyo, Japan
- Paul Stradins University Hospital, Riga, Latvia
- VU University Medical Center, Amsterdam, Netherlands
- Severance Cardiovascular Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rizvi A, Hartaigh BO, Knaapen P, Leipsic J, Shaw LJ, Andreini D, Pontone G, Raman S, Khan MA, Ridner M, Nabi F, Gimelli A, Jang J, Cole J, Nakazato R, Zarins C, Han D, Lee JH, Szymonifika J, Gomez MJ, Truong QA, Chang HJ, Lin FY, Min JK. Rationale and Design of the CREDENCE Trial: computed TomogRaphic evaluation of atherosclerotic DEtermiNants of myocardial IsChEmia. BMC Cardiovasc Disord. 2016 Oct 6;16(1):190. doi: 10.1186/s12872-016-0360-x. PMID 27716131
- [Derived] Lipkin I, Telluri A, Kim Y, Sidahmed A, Krepp JM, Choi BG, Jonas R, Marques H, Chang HJ, Choi JH, Doh JH, Her AY, Koo BK, Nam CW, Park HB, Shin SH, Cole J, Gimelli A, Khan MA, Lu B, Gao Y, Nabi F, Nakazato R, Schoepf UJ, Driessen RS, Bom MJ, Jang JJ, Ridner M, Rowan C, Avelar E, Genereux P, Knaapen P, de Waard GA, Pontone G, Andreini D, Al-Mallah MH, Crabtree TR, Earls JP, Choi AD, Min JK. Coronary CTA With AI-QCT Interpretation: Comparison With Myocardial Perfusion Imaging for Detection of Obstructive Stenosis Using Invasive Angiography as Reference Standard. AJR Am J Roentgenol. 2022 Sep;219(3):407-419. doi: 10.2214/AJR.21.27289. Epub 2022 Apr 20. PMID 35441530
- [Derived] Griffin WF, Choi AD, Riess JS, Marques H, Chang HJ, Choi JH, Doh JH, Her AY, Koo BK, Nam CW, Park HB, Shin SH, Cole J, Gimelli A, Khan MA, Lu B, Gao Y, Nabi F, Nakazato R, Schoepf UJ, Driessen RS, Bom MJ, Thompson R, Jang JJ, Ridner M, Rowan C, Avelar E, Genereux P, Knaapen P, de Waard GA, Pontone G, Andreini D, Earls JP. AI Evaluation of Stenosis on Coronary CTA, Comparison With Quantitative Coronary Angiography and Fractional Flow Reserve: A CREDENCE Trial Substudy. JACC Cardiovasc Imaging. 2023 Feb;16(2):193-205. doi: 10.1016/j.jcmg.2021.10.020. Epub 2022 Feb 16. PMID 35183478
- [Derived] Stuijfzand WJ, van Rosendael AR, Lin FY, Chang HJ, van den Hoogen IJ, Gianni U, Choi JH, Doh JH, Her AY, Koo BK, Nam CW, Park HB, Shin SH, Cole J, Gimelli A, Khan MA, Lu B, Gao Y, Nabi F, Nakazato R, Schoepf UJ, Driessen RS, Bom MJ, Thompson R, Jang JJ, Ridner M, Rowan C, Avelar E, Genereux P, Knaapen P, de Waard GA, Pontone G, Andreini D, Al-Mallah MH, Lu Y, Berman DS, Narula J, Min JK, Bax JJ, Shaw LJ; CREDENCE Investigators. Stress Myocardial Perfusion Imaging vs Coronary Computed Tomographic Angiography for Diagnosis of Invasive Vessel-Specific Coronary Physiology: Predictive Modeling Results From the Computed Tomographic Evaluation of Atherosclerotic Determinants of Myocardial Ischemia (CREDENCE) Trial. JAMA Cardiol. 2020 Dec 1;5(12):1338-1348. doi: 10.1001/jamacardio.2020.3409. PMID 32822476